CLINICAL TRIAL: NCT01216930
Title: Molecular Screening for Lynch Syndrome in Southern Denmark
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MS-LS-DK-01; 10-5156 (Other Grant/Funding Number: Region of Southern Denmark)
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer; Lynch Syndrome; HNPCC
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All colorectal cancer patients
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
A clinically applicably strategy for molecular screening for Lynch Syndrome has been implemented in the Region of Southern Denmark.

Based on sequential analysis with immunohistochemistry and methylation analysis, patients with possible hereditary colorectal cancer are identified. These patients are offered genetic risk assessment and counselling.

The study hypothesis is that molecular screening will identify more patients with Lynch Syndrome than the family history alone.

Prospective data collection is performed using established clinical databases.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of colorectal adenocarcinoma
* Diagnosed at one of the five departments of pathology in the region

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All colorectal cancer patients in the geographical region of southern Denmark
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Denmark (7):
  - Department of Pathology, Esbjerg
  - Department of Clinical Genetics, Odense
  - Department of Pathology, Odense
  - Department of Pahology, Svendborg
  - Department of Pathology, Sønderborg
  - Department of Clinical Genetics, Vejle
  - Department of Pathology, Vejle